CLINICAL TRIAL: NCT01226953
Title: A Phase III Observer Blind Single-Coordinating Center Pediatric Study in China Comparing a Booster Dose of Vaxem™ Hib to HIBERIX® When Given as Part of a Local Dosing Regimen in Infants
Brief Title: Immunogenicity and Safety of a Booster Dose of Monovalent Glycoprotein-Conjugated (Diptheria Toxin -CRM197) Hib Vaccine in 365-569 Days Old Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V37_07E1
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Haemophilus Influenzae Type b (Hib) Infection
Keywords: Haemophilus influenzae type b (Hib); Vaccine; Anti-PRP antibody
MeSH Terms: conditions — Haemophilus Infections; Infections | interventions — Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Biological: Haemophilus influenzae type b (Hib) vaccine
- Arm 2 (Active Comparator)
  Interventions: Biological: Haemophilus influenzae type b (Hib) vaccine

INTERVENTIONS:
Biological: Haemophilus influenzae type b (Hib) vaccine — Comparator study of two commercially available Haemophilus influenzae type b (Hib) vaccines

SUMMARY:
This study will evaluate the safety and immunogenicity of booster dose of two commercially available vaccines used to prevent Haemophilus influenzae type b infections in children 365-569 days of age

ELIGIBILITY:
Inclusion Criteria:

* Infants 365-569 days of age.

Exclusion Criteria:

* Subjects who already received a booster dose of Hib vaccine.
* History of serious reaction(s) following vaccination.
* Any vaccination within 7 days of study vaccination.
* Known or suspected immune impairment.

Ages: 365 Days to 569 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 660 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Anti-PRP (polyribosyl-ribitol-phosphate) antibody levels at day 31 post last vaccination | 30 days after last vaccination

SECONDARY OUTCOMES:
Solicited local and systemic reactions, adverse events (AEs), and serious adverse events (SAEs) | 30 days post last vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Province, China

REFERENCES:
- [Derived] Jun L, Yuguo C, Zhiguo W, Jinfeng L, Huawei M, Xiuhua L, Yonggui Z, Yanhua X, Kong Y, Hongtao L, Yuliang Z. Assessment of immunogenicity and safety following primary and booster immunisation with a CRM197 -conjugated Haemophilus influenzae type B vaccine in healthy Chinese infants. Int J Clin Pract. 2013 Oct;67(10):971-8. doi: 10.1111/ijcp.12267. Epub 2013 Aug 22. PMID 23964690